CLINICAL TRIAL: NCT04220996
Title: Interventional, Open-label Effectiveness Study of Flexible Doses of Vortioxetine on Depressive Symptoms in Patients With Major Depressive Disorder Comorbid With Generalized Anxiety Disorder
Brief Title: Vortioxetine in Patients With Depression Coexisting With General Anxiety Disorder (GAD)
Acronym: RECONNECT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18314A
Record Dates: First submitted 2020-01-06; First posted 2020-01-07 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: MDD; Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders | interventions — Vortioxetine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vortioxetine (Experimental): 10-20 mg vortioxetine tablets
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — Vortioxetine 10 and 20 mg/day, tablets, orally Patients will receive 10 mg vortioxetine once daily for the first week. At Visit 2, the dose will be increased to 20 mg/day. The dose may subsequently be adjusted to 10 or 20 mg/day at scheduled or unscheduled visits depending on patient's response as per investigator judgment.

SUMMARY:
This study evaluates the effectiveness of vortioxetine on depressive symptoms in patients with depression coexisting with generalized anxiety disorder.

DETAILED DESCRIPTION:
100 patients, recruited from psychiatrist outpatient clinics are planned for enrolment. Approximately 50 of these patients will receive vortioxetine as a first treatment for the current Major Depressive Episode (MDE) (first treatment patients) and 50 patients will be switched to vortioxetine due to inadequate response to the current antidepressant medication treatment (switch patients).

ELIGIBILITY:
Inclusion Criteria:

* The patient has a primary diagnosis of MDE, diagnosed according to DSM-5® confirmed using the Mini International Neuropsychiatric Interview (MINI).
* The patient has had the current MDE for <12 months
* The patient has current comorbid Generalized Anxiety Disorder (GAD) according to DSM-5®. The diagnosis was made prior to the current MDE
* The patient has a Montgomery and Åsberg Depression Rating Scale (MADRS) total score ≥ 22 at the Baseline Visit
* The patient has a Hamilton Anxiety Rating Scale (HAM-A) score ≥ 20 at the Baseline Visit

Exclusion Criteria:

* The patient has any current psychiatric disorder or Axis I disorder (DSM-5® criteria), established as the primary diagnosis, other than MDD, as assessed using the Mini International Neuropsychiatric Interview (MINI) or another diagnostic interview.
* The patient has a history of previous major depressive episodes considered as treatment resistant, defined as inadequate response (incomplete or no therapeutic response) to two prior courses of at least 6 weeks of conventional antidepressant drugs in adequate dosages or, the patient has treatment-resistant depression in the investigator's opinion.

Other in- or exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-12-27 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-03-09 (Actual)

PRIMARY OUTCOMES:
Change in Montgomery and Åsberg Depression Rating Scale (MADRS) total score | from baseline to Week 8
  The Montgomery and Åsberg Depression Rating Scale (MADRS) is a 10-item rating scale designed to assess the severity of the symptoms in depressive illness and to be sensitive to treatment effects. Symptoms are rated on a 7-point scale from 0 (no symptom) to 6 (severe symptom). The total score of the 10 items ranges from 0 to 60, with higher values indicating worse outcome.

SECONDARY OUTCOMES:
Change in Hamilton Anxiety Rating Scale (HAM-A) total score | from baseline to Week 8
  The HAM-A is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 to 56 where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. Total scores above 30 indicate very severe anxiety.
Change in Hospital Anxiety and Depression Scale (HADS) total score | from baseline to Week 8
  The HADS is a patient-rated scale designed to screen for anxiety and depressive states in medical patients. It consists of two sub-scales: the D-scale measures depression and the A-scale measures anxiety. Each sub-scale contains 7 items, and each item is rated from 0 (absent) to 3 (maximum severity). The score of each sub-scale ranges from 0 to 21.
Change in Functioning Assessment Short Test (FAST) total score | from baseline to Week 8
  The FAST is a valid and reliable instrument, easy to apply which requires a short period of time to administer. Evaluates functioning taking into account the last 15 days. It was developed for the clinical evaluation of the main difficulties presented by psychiatric patients, and has been validated in several languages for patients with bipolar disorder. The FAST scale consists of 24 items which allow the assessment of six specific areas of functioning: autonomy, occupational functioning, cognitive functioning, financial issues, interpersonal relationships and leisure time. Each item is rated on a 4-point scale from 0 (no difficulty) to 3 (severe difficulty). The items are summed to yield a total score ranging from 0 to 72 with higher scores reflecting more serious difficulties.
Change in Clinical Global Impression - Severity of Illness (CGI-S) score | from baseline to Week 8
  The Clinical Global Impression severity of illness (CGI-S) provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (normal - not at all ill) to 7 (among the most extremely ill patients).
Clinical Global Impression Scale- Global Improvement (CGI-I) score | At Week 8
  The Clinical Global Impression - global improvement CGI-I provides the clinician's impression of the patient's improvement (or worsening). The clinician assesses the patient's condition relative to a baseline on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse).
Change in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) total score | from baseline to Week 8
  The original Q-LES-Q is a patient self-rated scale designed to measure the degree of enjoyment and satisfaction experienced by patients in various areas of daily life. It consists of 93 items to measure: physical health, feelings, work, household duties, school, leisure time activities, social relations, and general activities. Each item is rated on a 5-point scale ranging from 1 (very poor) to 5 (very good).

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (21):
- Estonia (2):
  - Marienthali Kliinik (EE0001), Tallinn
  - Tartu University Hospital (EE0002), Tartu
- France (4):
  - Cabinet du Docteur Patrick Bourgoin (FR0002), Angoulême
  - Cabinet Psyche (FR0004), Douai
  - Centre Medical Ambroise Pare (FR0003), Élancourt
  - Cabinet du Docteur Karim Boutayeb (FR0001), Viersat
- Italy (2):
  - Azienda Ospedaliera di Perugia - Policlinico Monteluce (IT0003), Perugia
  - Fondazione Santa Lucia IRCCS (IT0002), Rome
- Poland (8):
  - MlynowaMed Specjalistyczny Psychiatryczny Gabinet Lekarski Joanna Lazarczyk (PL0009), Bialystok
  - NZOZ Dom Sue Ryder - Pallmed Sp. z o.o. (PL0003), Bydgoszcz
  - CareClinic (PL0005), Katowice
  - Centrum Zdrowia Psychicznego Biomed - Jan Latala (PL0001), Kielce
  - Niepubliczny Zaklad Opieki Psychiatrycznej Mentis (PL0004), Leszno
  - Centrum Medyczne Luxmed Sp.Z O.O. (PL0006), Lublin
  - Clinical Research Center Spolka z ograniczona odpowiedzialnoscia Medic-R Sp.k. (PL0007), Poznan
  - Nzoz Syntonia (PL0010), Pruszcz Gdański
- South Korea (3):
  - Inje University Ilsan Paik Hospital (KR0002), Goyang-si
  - Chonnam National University Hospital (KR0003), Gwangju
  - Samsung Medical Center (KR0001), Seoul
- Spain (2):
  - Hospital Clinic de Barcelona (ES0003), Barcelona
  - Instituto Internacional de Neurociencias Aplicadas (ES0001), Barcelona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Christensen MC, Schmidt S, Grande I. Effectiveness of vortioxetine in patients with major depressive disorder comorbid with generalized anxiety disorder: Results of the RECONNECT study. J Psychopharmacol. 2022 May;36(5):566-577. doi: 10.1177/02698811221090627. Epub 2022 May 2. PMID 35499104